CLINICAL TRIAL: NCT06444347
Title: The Impact of Biosynthetic Mesh on Paraesophageal Hernia Repair in Robotic Anti-Reflux Surgery: A Multi-Institutional Randomized Trial
Brief Title: Impact of Biosynthetic Mesh on Paraesophageal Hernia Repair
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-11026766
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Hiatal Hernia
MeSH Terms: conditions — Hernia, Hiatal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Biosynthetic Mesh (Experimental): The biosynthetic mesh group will undergo hiatal hernia repair with Phasix Mesh (Becton Dickinson, Franklin Lakes, NJ) reinforcement, secured with permanent suture. This is a biosynthetic mesh that completely reabsorbs in 12-18 months after surgery. The mesh is designed to provide strength during the initial healing phase after hernia repair, allowing for rapid tissue ingrowth and vascularization, gradually transferring the load to native tissue as it resorbs1. This mesh has been FDA approved for procedures involving soft tissue repair, such as hernia defects.
  Interventions: Device: Biosynthetic Mesh; Procedure: Hiatal Hernia Repair
- No Mesh (Active Comparator): The non-mesh group will undergo repair with permanent suture only.
  Interventions: Procedure: Hiatal Hernia Repair

INTERVENTIONS:
Device: Biosynthetic Mesh — The biosynthetic mesh group will undergo hiatal hernia repair with Phasix Mesh (Becton Dickinson, Franklin Lakes, NJ) reinforcement, secured with permanent suture.
  Arms: Biosynthetic Mesh
Procedure: Hiatal Hernia Repair — The non-mesh group will undergo hiatal hernia repair with permanent suture only.

SUMMARY:
The aim of this study is to find out if using a certain kind of mesh can reduce the chances of hiatal hernias coming back after anti-reflux surgery. Participants undergoing antireflux surgery will be assigned to one of two groups, a group that has surgery with mesh, or a group that has surgery without mesh.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of gastroesophageal reflux disease
* Adults aged 18 years or older
* English speaking
* Subject is planned to undergo surgery for reflux disease

Exclusion Criteria:

* Physician deems the subject is unable to complete the study due to documented dementia.
* Subject is undergoing emergent surgery.
* Pregnancy
* Patient has known allergy to tetracycline hydrochloride or kanamycin sulfate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Anatomic hiatal hernia recurrence rate | 1 year

SECONDARY OUTCOMES:
Anatomic Hiatal Hernia Recurrence rate | 3 years
Anatomic Hiatal Hernia Recurrence rate | 5 years
Reflux Symptoms | 2 weeks postoperatively
  Reflux symptoms will be assessed using the gastroesophageal reflux disease health related quality of life survey (GERD-HRQL). The highest possible score on this survey is 75, indicating daily incapacitating symptoms in all areas assessed. The lowest possible score is 0, indicating no symptoms.
Reflux Symptoms | 6 months postoperatively
  Reflux symptoms will be assessed using the gastroesophageal reflux disease health related quality of life survey (GERD-HRQL). The highest possible score on this survey is 75, indicating daily incapacitating symptoms in all areas assessed. The lowest possible score is 0, indicating no symptoms.
Reflux Symptoms | 1 year postoperatively
  Reflux symptoms will be assessed using the gastroesophageal reflux disease health related quality of life survey (GERD-HRQL). The highest possible score on this survey is 75, indicating daily incapacitating symptoms in all areas assessed. The lowest possible score is 0, indicating no symptoms.
Reflux Symptoms | 2 years postoperatively
  Reflux symptoms will be assessed using the gastroesophageal reflux disease health related quality of life survey (GERD-HRQL). The highest possible score on this survey is 75, indicating daily incapacitating symptoms in all areas assessed. The lowest possible score is 0, indicating no symptoms.
Reflux Symptoms | 3 years postoperatively
  Reflux symptoms will be assessed using the gastroesophageal reflux disease health related quality of life survey (GERD-HRQL). The highest possible score on this survey is 75, indicating daily incapacitating symptoms in all areas assessed. The lowest possible score is 0, indicating no symptoms.
Reflux Symptoms | 4 years postoperatively
  Reflux symptoms will be assessed using the gastroesophageal reflux disease health related quality of life survey (GERD-HRQL). The highest possible score on this survey is 75, indicating daily incapacitating symptoms in all areas assessed. The lowest possible score is 0, indicating no symptoms.
Reflux Symptoms | 5 years postoperatively
  Reflux symptoms will be assessed using the gastroesophageal reflux disease health related quality of life survey (GERD-HRQL). The highest possible score on this survey is 75, indicating daily incapacitating symptoms in all areas assessed. The lowest possible score is 0, indicating no symptoms.
Dysphagia Symptoms | 2 weeks postoperatively
  Dysphagia symptoms will be assessed using the Bazaz dysphagia score. The lowest dysphagia severity score being "none", indicating no difficulty swallowing. The highest dysphagia severity score being "severe", indicating frequent difficulty swallowing with the majority of foods.
Dysphagia Symptoms | 6 months postoperatively
  Dysphagia symptoms will be assessed using the Bazaz dysphagia score. The lowest dysphagia severity score being "none", indicating no difficulty swallowing. The highest dysphagia severity score being "severe", indicating frequent difficulty swallowing with the majority of foods.
Dysphagia Symptoms | 1 year postoperatively
  Dysphagia symptoms will be assessed using the Bazaz dysphagia score. The lowest dysphagia severity score being "none", indicating no difficulty swallowing. The highest dysphagia severity score being "severe", indicating frequent difficulty swallowing with the majority of foods.
Dysphagia Symptoms | 2 years postoperatively
  Dysphagia symptoms will be assessed using the Bazaz dysphagia score. The lowest dysphagia severity score being "none", indicating no difficulty swallowing. The highest dysphagia severity score being "severe", indicating frequent difficulty swallowing with the majority of foods.
Dysphagia Symptoms | 3 years postoperatively
  Dysphagia symptoms will be assessed using the Bazaz dysphagia score. The lowest dysphagia severity score being "none", indicating no difficulty swallowing. The highest dysphagia severity score being "severe", indicating frequent difficulty swallowing with the majority of foods.
Dysphagia Symptoms | 4 years postoperatively
  Dysphagia symptoms will be assessed using the Bazaz dysphagia score. The lowest dysphagia severity score being "none", indicating no difficulty swallowing. The highest dysphagia severity score being "severe", indicating frequent difficulty swallowing with the majority of foods.
Dysphagia Symptoms | 5 years postoperatively
  Dysphagia symptoms will be assessed using the Bazaz dysphagia score. The lowest dysphagia severity score being "none", indicating no difficulty swallowing. The highest dysphagia severity score being "severe", indicating frequent difficulty swallowing with the majority of foods.
Number of subjects requiring 30 day readmission | 30 days following surgery
Number of subjects requiring reoperation | 30 days following surgery
Number of subjects developing postoperative Infection | 30 days following surgery

CONTACTS AND LOCATIONS:
Overall Officials: Rasa Zarnegar, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (6):
- United States (6):
  - University of Southern California Keck School of Medicine, Los Angeles, California
  - Louisiana State University School of Medicine, New Orleans, Louisiana
  - Washington University School of Medicine, St Louis, Missouri
  - NYU Langone Health, New York, New York
  - Weill Cornell Medicine, New York, New York
  - Lenox Hill Hospital, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yamasaki T, Hemond C, Eisa M, Ganocy S, Fass R. The Changing Epidemiology of Gastroesophageal Reflux Disease: Are Patients Getting Younger? J Neurogastroenterol Motil. 2018 Oct 1;24(4):559-569. doi: 10.5056/jnm18140. PMID 30347935
- [Background] Li Q, Blume SW, Huang JC, Hammer M, Ganz ML. Prevalence and healthcare costs of obesity-related comorbidities: evidence from an electronic medical records system in the United States. J Med Econ. 2015;18(12):1020-8. doi: 10.3111/13696998.2015.1067623. Epub 2015 Sep 4. PMID 26134917
- [Background] Oelschlager BK, Pellegrini CA, Hunter JG, Brunt ML, Soper NJ, Sheppard BC, Polissar NL, Neradilek MB, Mitsumori LM, Rohrmann CA, Swanstrom LL. Biologic prosthesis to prevent recurrence after laparoscopic paraesophageal hernia repair: long-term follow-up from a multicenter, prospective, randomized trial. J Am Coll Surg. 2011 Oct;213(4):461-8. doi: 10.1016/j.jamcollsurg.2011.05.017. Epub 2011 Jun 29. PMID 21715189
- [Background] Spiro C, Quarmby N, Gananadha S. Mesh-related complications in paraoesophageal repair: a systematic review. Surg Endosc. 2020 Oct;34(10):4257-4280. doi: 10.1007/s00464-020-07723-0. Epub 2020 Jun 18. PMID 32556700
- [Background] Deeken CR, Matthews BD. Characterization of the Mechanical Strength, Resorption Properties, and Histologic Characteristics of a Fully Absorbable Material (Poly-4-hydroxybutyrate-PHASIX Mesh) in a Porcine Model of Hernia Repair. ISRN Surg. 2013 May 28;2013:238067. doi: 10.1155/2013/238067. Print 2013. PMID 23781348
- [Background] Alicuben ET, Worrell SG, DeMeester SR. Resorbable biosynthetic mesh for crural reinforcement during hiatal hernia repair. Am Surg. 2014 Oct;80(10):1030-3. PMID 25264654
- [Background] Aiolfi A, Cavalli M, Sozzi A, Lombardo F, Lanzaro A, Panizzo V, Bonitta G, Mendogni P, Bruni PG, Campanelli G, Bona D. Medium-term safety and efficacy profile of paraesophageal hernia repair with Phasix-ST(R) mesh: a single-institution experience. Hernia. 2022 Feb;26(1):279-286. doi: 10.1007/s10029-021-02528-z. Epub 2021 Oct 30. PMID 34716832
- [Background] Tartaglia E, Cuccurullo D, Guerriero L, Reggio S, Sagnelli C, Mugione P, Corcione F. The use of biosynthetic mesh in giant hiatal hernia repair: is there a rationale? A 3-year single-center experience. Hernia. 2021 Oct;25(5):1355-1361. doi: 10.1007/s10029-020-02273-9. Epub 2020 Jul 25. PMID 32712835
- [Background] Panici Tonucci T, Asti E, Sironi A, Ferrari D, Bonavina L. Safety and Efficacy of Crura Augmentation with Phasix ST Mesh for Large Hiatal Hernia: 3-Year Single-Center Experience. J Laparoendosc Adv Surg Tech A. 2020 Apr;30(4):369-372. doi: 10.1089/lap.2019.0726. Epub 2020 Jan 7. PMID 31910348
- [Background] Quake, S. Y. L., Peter, B., Munipalle, P. C., & Viswanath, Y. (2023). OGBN O08 The Safety and Efficacy of Laparoscopic Hiatus Hernia Repair with Biosynthetic Mesh (Phasix-ST®): A Single Centre Experience. British Journal of Surgery, 110(Supplement_8), znad348-030.
- [Background] Konstantinidis H, Charisis C. Surgical treatment of large and complicated hiatal hernias with the new resorbable mesh with hydrogel barrier (Phasix ST): a preliminary study. J Robot Surg. 2023 Feb;17(1):141-146. doi: 10.1007/s11701-022-01406-9. Epub 2022 Apr 9. PMID 35397107
- [Background] Abdelmoaty WF, Dunst CM, Filicori F, Zihni AM, Davila-Bradley D, Reavis KM, Swanstrom LL, DeMeester SR. Combination of Surgical Technique and Bioresorbable Mesh Reinforcement of the Crural Repair Leads to Low Early Hernia Recurrence Rates with Laparoscopic Paraesophageal Hernia Repair. J Gastrointest Surg. 2020 Jul;24(7):1477-1481. doi: 10.1007/s11605-019-04358-y. Epub 2019 Aug 29. PMID 31468330
- See also: "PhasixTM Mesh." — https://www.bd.com/en-us/products-and-solutions/products/product-families/phasix-mesh.